CLINICAL TRIAL: NCT04107974
Title: Percutaneous Radiologic Gastrostomy With and Without Gastropexy: A Prospective Comparison
Brief Title: PRG With and Without Gastropexy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ganesan Annamalai, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-5102
Record Dates: First submitted 2019-05-20; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Gastrostomy; Gastrostomy Complications
Keywords: Gastropexy; Percutaneous Radiologic Gastrostomy; Interventional Radiology
MeSH Terms: interventions — Gastropexy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing gastropexy to non-gastropexy for quality of life and complications.
Who Masked: Outcomes Assessor
Masking Description: Patients and interventional radiologists cannot be blinded to the procedure as the follow up and performing the procedure for gastropexy versus non-gastropexy is different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gastropexy (Experimental): Percutaneous radiologic guided insertion of G-tube. The skin over the epigastrium is prepared and draped in sterile fashion. Midazolam and fentanyl are administered for conscious sedation. Lidocaine for local analgesia. The stomach is insufflated with air after insertion of an OG or NG tube. Two T-fasteners are inserted into the stomach approximately 4cm apart. A needle is inserted into the stomach and an Amplatz wire is then inserted into the stomach. The tract is dilated with an 18Fr peel away sheath. A 14 Fr balloon retention gastrostomy tube is inserted. The balloon is inflated and bolster set as appropriate. The gastropexy/T-fastener sutures are cut after one week.
  Interventions: Device: Gastropexy.
- Non-Gastropexy (Experimental): Percutaneous radiologic guided insertion of G-tube. The skin over the epigastrium is prepared and draped in sterile fashion. Midazolam and fentanyl are administered for conscious sedation. Lidocaine for local analgesia. The stomach is insufflated with air after insertion of an OG or NG tube. A needle is inserted into the stomach and an Amplatz wire is then inserted into the stomach. The tract is dilated with an 18Fr peel away sheath. A 14 Fr balloon retention gastrostomy tube is inserted. The balloon is inflated and bolster set as appropriate.
  Interventions: Procedure: Non-Gastropexy

INTERVENTIONS:
Device: Gastropexy. — Two T-fasteners for G-tube insertion (gastropexy).
  Arms: Gastropexy
Procedure: Non-Gastropexy — Insertion of G-tube in absence of T-fasteners.
  Arms: Non-Gastropexy

SUMMARY:
Percutaneous (through the skin) radiologic (x-ray guided) gastrostomy (to the stomach) (PRG) is a common procedure performed to help provide supplemental nutrition for those for who have difficulty swallowing their food. This population typically includes patients receiving radiation therapy for cancers of the mouth or throat, patients who have had a stroke or other neurologic disorders. It involves making a small incision in the skin on the belly to insert a feeding tube directly into the stomach. PRG has been well established as a safe and effective procedure for many years now. Although known to be safe, there is still debate regarding the best way to perform the procedure. Some doctors believe it is necessary to stitch the stomach wall against the wall of the belly before inserting the tube, this is called gastropexy. They argue that this decreases the risk of the tube being positioned incorrectly and prevents leakage of stomach content in the first few weeks after the procedure. Other doctors feel that these risks are very small and this step is not required as it can cause the patient more pain in the days following the procedure since the stomach is fixed against the body wall and cannot move naturally. To this day, the procedure is performed safely both ways, depending on the hospital.

The purpose of this research study is to compare these two methods and determine if one technique gives better results, meaning less pain and fewer complications for patients.

DETAILED DESCRIPTION:
When percutaneous radiological gastrostomy (PRG) first emerged as an alternative method to surgical or endoscopic techniques, gastropexy was considered an essential step. This consists of using sutures and "T-fasteners" to fix the anterior gastric wall to the anterior abdominal wall and many variations are described in the literature. It was postulated that this step is necessary to avoid tube misplacement and peritonitis caused by early leakage of gastric content around the site of tube insertion. It is still considered imperative in some groups of patients at high risk of gastric leakage (i.e. patients with ascites, steroid treatment, and/or severe malnourishment). However, in other patients its use has become subject of debate.

Experiments with animal models have shown no evidence of gastric leakage following insertion of a 14 French tube, even when the tube is subsequently removed and the defect left unrepaired. Furthermore, several groups have had success without the use of gastropexy and some have described complications caused by performing this step such as peristomal infection, increased post-procedural pain, persistent leakage, and gastrocutaneous fistulas. Other large series of patients who underwent gastrostomy with gastropexy did not experience gastropexy-related complications, further complicating the matter. To date, the guidelines for transabdominal gastrostomy published by the Society of Interventional Radiology (SIR) and American Gastroenterological Association (AGA) acknowledge both techniques but have no official recommendation on the use of gastropexy reflecting the lack of clear evidence regarding advantage with or without its use.

The investigators hypothesize that the use of gastropexy for PRG does not significantly decrease complications.

The investigators also hypothesize that the use of gastropexy is associated with increased post procedural pain.

At the investigators' institution (University Health Network) PRG without gastropexy is regularly performed first-line for gastrostomy. There is a high volume of requests for PRG and thus establishing which method is superior will help to reduce the number of complications and revisions. In doing so, the investigators hope to be able to establish an optimal evidence-based protocol for PRG for future patients as well as improving patient safety and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years and older) meeting standard eligibility criteria for percutaneous radiologic gastrostomy
* Dysphagia related to malignancy or surgery/radiation therapy
* Able to appropriately understand and complete English questionnaires either independently or with the assistance of a translator

Exclusion Criteria:

* Unable to provide informed consent
* Unable or unwilling to complete the pre and post-procedure questionnaires
* Dysphagia related to neurological deficits
* Large volume of ascites
* Prior partial gastrectomy
* Long-term steroid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-11 (Estimated); Study Completion 2019-11-11 (Estimated)

PRIMARY OUTCOMES:
Pain level as reported on 10-point Visual Analog Scale | Pre-procedure baseline measure, post-procedure (day 1) measure, and 30 day post-procedure measure
  10-point Visual Analog Scale (VAS) (0 = no pain, 10 = worst pain imaginable) with specific procedure-related questions, as outlined in the pre- and post-procedure questionnaire.

SECONDARY OUTCOMES:
Complications | 30 days post-procedure follow-up.
  Number of participants who experienced procedure-related complications (major and minor) in each arm will be assessed according to established criteria (ie SIR Adverse Event Classification).

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a single center trial. Only researchers at this site will have access to the participant data.